CLINICAL TRIAL: NCT07075510
Title: A Phase I/II Study of Subcutaneous Daratumumab Administration in the Anterior Upper Thigh Vs Abdomen in Patients With Plasma Cell Disorders
Brief Title: Subcutaneous Daratumumab Administration in the Thigh Vs Abdomen in Plasma Cell Disorders
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2513GCCC; HP-00113670 (Other: UMB IRB)
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Plasma Cell Disorder
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ArmA: Treatment with Subcutaneous Daratumumab Administration in the Anterior Upper Thigh (Experimental): Treatment will be given for 8 weeks. SC Daratumumab will be administered in the thigh weekly for 8 weeks. Patients may receive daratumumab alone or in combination with standard of care regimen
  Interventions: Drug: Daratumumab Injection
- ArmB: Treatment with Subcutaneous Daratumumab Administration in the Abdomen (Active Comparator): Treatment will be given for 8 weeks. SC Daratumumab will be administered in the abdomen weekly for 8 weeks. Patients may receive daratumumab alone or in combination with standard of care regimen
  Interventions: Drug: Daratumumab Injection

INTERVENTIONS:
Drug: Daratumumab Injection — Daratumumab Administration in the Anterior Upper Thigh versus the Abdomen

SUMMARY:
The purpose of this study is to look at the safety, tolerability, and serum concentration of daratumumab administered subcutaneously in the thigh versus the abdomen in patients with plasma cell disorders. Daratumumab is a monoclonal antibody that can attach itself to the CD38 protein on the surface of abnormal plasma cells. Daratumumab can kill the abnormal plasma cells and/or help your immune system find and destroy them. Due to the way daratumumab works, normal cells may also be affected. All reference to the words "study drug" in this consent form will mean Daratumumab.

Daratumumab has been approved by the U.S. Food and Drug Administration (FDA) alone or in combination with other standard of care drugs for treatment of multiple myeloma in both subcutaneous (DARZALEX FASPRO®) and intravenous (DARZALEX®) ways of being delivered. The FDA has also approved the subcutaneous administration of daratumumab combined with other standard of care drugs for patients with light chain (AL) amyloidosis. Subcutaneous means the drug is given by an injection just beneath the skin. Intravenous (IV) means the drug is given as an injection directly into a vein.

Usually when given subcutaneously, the study drug is given by an injection in the abdomen. Having the drug given by subcutaneous injection (underneath the skin of the abdomen) has lessened the IV related side effects and the drug administration by injection is quicker.

However, some patients cannot receive the study drug injections in their abdomen because they find them very painful or have other medical reasons making it difficult to get these injections. The goal of this study is to see if getting the study drug subcutaneously, injected under the skin by a needle, in the patient's upper thigh will have the same results, or better results, as getting the injection in the abdomen. This would therefore, improve patients access to the drug and provide an alternative place to receive the injection of the drug.

This study will take place at University of Maryland Medical Center and there will be about 30 people who will take place in this study here. Dr. Badros is the Sponsor-Investigator of the study. Funding to conduct the study and study drug are being provided by Johnson & Johnson Innovative Medicine (J&J IM).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of MM (newly diagnosed or relapsed) or AL amyloid with planned therapy with daratumumab-based regimen. and has not received daratumumab previously or has received daratumumab > 6 months prior to planned Cycle 1 Day 1 alone or in combination with other regimens per investigator discretion.
2. Provide signed written informed consent
3. 18 years or older (at the time consent is obtained)
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
5. Participants with a history of autologous stem cell transplant or prior CAR-T cell therapy can enroll on the study provided that:

   1. Therapy was >100 days prior to study enrollment
   2. No active infection(s)
6. Adequate organ system function
7. Female participants: Contraceptive use for those participating in clinical studies (men or women) should be consistent with local regulations: A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

   1. Is not a woman of childbearing potential (WOCBP) OR
   2. Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, during the intervention period and for at least 12 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The Investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

      * A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study intervention.
      * We will review the medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a new undetected pregnancy.

   Non childbearing potential is defined as follows (by other than medical reasons):
   * ≥45 years of age and has not had menses for >1 year
   * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range
   * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation.
8. Male participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Male participants are eligible to participate if they agree to the following during the intervention period and for 6 months after the last dose of study treatment to allow for clearance of any altered sperm:

   a. Refrain from donating sperm PLUS either:
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent. OR
   * Must agree to use contraception/barrier and use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse with a woman of childbearing potential
9. All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0) must be ≤ Grade 1 at the time of enrollment except for alopecia and Grade 2 peripheral neuropathy.
10. Participants are able to comply with visit schedule and agree to weekly visits for 9 weeks

Exclusion Criteria:

1. Systemic anti-myeloma therapy within ≤14 days or 5 half-lives, whichever is shorter, or plasmapheresis within 7 days prior to the first dose of study drug
2. Systemic treatment with high dose steroids (equivalent to >60 mg prednisone daily for ≥4 days) within the past 14 days if administered to treat MM or non- MM disease
3. Evidence of active bleeding
4. Any major surgery within the last 28 days
5. Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided participants fulfil entry criteria (as defined by inclusion criteria #6)
6. Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere participants' safety, obtaining informed consent or compliance with study procedures.
7. Current unstable liver disease per Investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. NOTE: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) is acceptable if participant otherwise meets entry criteria.
8. Other malignancies are excluded, except for malignancy from which the patients have been disease-free for more than 2 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, prostate cancer or in situ cervical or breast cancer that has undergone potentially curative therapy.
9. Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is < 50% of predicted normal.
10. Moderate or severe persistent asthma within the past 2 years (see Attachment XX), or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate.
11. History of cardiovascular disease including any of the following:

    1. History of clinically significant untreated arrhythmias, including clinically significant ECG abnormalities including second degree (Mobitz Type II) or third degree atrioventricular (AV) block.
    2. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of screening.
    3. Class III or IV heart failure as defined by the New York Heart Association functional classification system.
    4. Uncontrolled hypertension.
12. Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to daratumumab
13. Active infection requiring treatment.
14. Presence of hepatitis B surface antigen (HbsAg), or hepatitis B core antibody (HbcAb), at screening or within 3 months prior to first dose of study treatment. Note: presence of Hep B surface antibody positivity as the only serologic marker (HBsAb) indicating previous vaccination will not exclude a participant provided that patient has a known history of prior HBV vaccination Positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment. NOTE: Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained. Hepatitis RNA testing is optional and participants with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing.
15. Pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Time of first dose (week 1), up to 8 doses (week 9)
  To characterize the safety and tolerability of subcutaneous daratumumab administered in the thigh vs the abdomen in patients with plasma cell disorders.
  Frequency and incidence rate of adverse events by type, severity, timing, and attribution to study drug, according to the NCI-CTCAE version 5.0.

SECONDARY OUTCOMES:
Measure of maximum serum trough concentration of daratumumab [Pharmacokinetic (PK) Analysis] | Time of first dose (week 1), up to 8 doses (week 9)
  To assess serum concentrations of daratumumab administered in the thigh vs the abdomen in patients with plasma cell disorders.
  To measure maximum serum trough concentration of daratumumab, defined as the pre-dose serum concentration of daratumumab on Week 9, Day 1 (after 8 weekly doses)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Badros, MD, Principal Investigator — University of Maryland, Baltimore Greenebaum Comprehensive Cancer Center
Locations (1):
- University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mateos MV, Nahi H, Legiec W, Grosicki S, Vorobyev V, Spicka I, Hungria V, Korenkova S, Bahlis N, Flogegard M, Blade J, Moreau P, Kaiser M, Iida S, Laubach J, Magen H, Cavo M, Hulin C, White D, De Stefano V, Clemens PL, Masterson T, Lantz K, O'Rourke L, Heuck C, Qin X, Parasrampuria DA, Yuan Z, Xu S, Qi M, Usmani SZ. Subcutaneous versus intravenous daratumumab in patients with relapsed or refractory multiple myeloma (COLUMBA): a multicentre, open-label, non-inferiority, randomised, phase 3 trial. Lancet Haematol. 2020 May;7(5):e370-e380. doi: 10.1016/S2352-3026(20)30070-3. Epub 2020 Mar 23. PMID 32213342
- [Background] Mateos M-V, Usmani SZ, Grosicki S, et al. Randomized, Open-Label, Non-Inferiority, Phase 3 Study of Subcutaneous (SC) Versus Intravenous (IV) Daratumumab (DARA) Administration in Patients (Pts) with Relapsed or Refractory Multiple Myeloma (RRMM): Body Weight Subgroup Analysis of Columba. Blood. 2019;134(Supplement 1):1906. doi:10.1182/blood-2019-122501
- [Background] Usmani SZ, Mateos M-V, Nahi H, et al. Randomized, Open-Label, Non-Inferiority, Phase 3 Study of Subcutaneous (SC) Versus Intravenous (IV) Daratumumab (DARA) Administration in Patients with Relapsed or Refractory Multiple Myeloma: Columba Update. Blood. 2019;134(Supplement 1):1865. doi:10.1182/blood-2019- 122765
- [Background] Zou P, Wang F, Wang J, Lu Y, Tran D, Seo SK. Impact of injection sites on clinical pharmacokinetics of subcutaneously administered peptides and proteins. J Control Release. 2021 Aug 10;336:310-321. doi: 10.1016/j.jconrel.2021.06.038. Epub 2021 Jun 26. PMID 34186147
- [Background] Reinisch M, Untch M, Mahlberg R, Reimer T, Hitschold T, Marme F, Aydogdu M, Schmatloch S, Luck HJ, Schmidt M, Ladda E, Sinn BV, Klare P, Janni W, Jackisch C, Denkert C, Seiler S, Gohler T, Michel L, Burchardi N, Stickeler E, Rey J, Klutinus N, Mobus V, Loibl S. Subcutaneous injection of trastuzumab into the thigh versus abdominal wall in patients with HER2-positive early breast cancer: Pharmacokinetic, safety and patients' preference - Substudy of the randomised phase III GAIN-2 study. Breast. 2022 Dec;66:110-117. doi: 10.1016/j.breast.2022.10.002. Epub 2022 Oct 5. PMID 36223695
- See also: Related Info — https://www.janssenlabels.com/package-insert/product-monograph/prescribing-information/DARZALEX+Faspro-pi.pdf